CLINICAL TRIAL: NCT06780488
Title: Visuo-Vestibular VR-based Stimulation Effects on Balance and Gait in Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 171/SL/24
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Stroke
Keywords: Stroke; Vestibular Rehabilitation; Virtual Reality; Balance; Gait; Quality of Life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real (Experimental)
  Interventions: Other: Real Visual-Vestibuar Rehabilitation
- Control (Sham Comparator)
  Interventions: Other: Sham Rehabilitation

INTERVENTIONS:
Other: Real Visual-Vestibuar Rehabilitation — The "Real Visual-Vestibular Rehabilitation" protocol will consist of specific exercises aimed at stimulating the visuo-vestibular function within immersive virtual reality environments replicating daily life situations. Patients will perform exercises in two types of contexts. In all exercises, patients will be free to move within a room large enough to complete the tasks. Walking during the exercises can also be performed with assistive devices, to make the context as close as possible to the patient's daily life. During the exercises, patients will be supervised by a physiotherapist specialized in neurological and vestibular rehabilitation.The protocol will last 20 minutes, with 10 minutes dedicated to each exercise.
  Arms: Real
Other: Sham Rehabilitation — The "Sham Vestibular Rehabilitation" protocol will involve the use of the same immersive virtual reality contexts and will aim to achieve the same objectives as the Real Visual-Vestibular Rehabilitation protocol, but without the "unexpected" stimuli. In both exercises, patients will be free to move within a room large enough to complete the tasks. Walking during the session can also be performed with assistive devices, to make the context as close as possible to the patient's daily life. During the exercises, patients will be supervised by a physiotherapist specialized in neurological and vestibular rehabilitation. The protocol will last 20 minutes, with 10 minutes dedicated to each exercise.
  Arms: Control

SUMMARY:
This pilot study aims to evaluate the effect of a specfic Virtual-Reality-Based rehabilitation training in patients with stroke. A total of 38 patients with stroke (more than 6 months from the acute event), recruited from the services of the Fondazione Santa Lucia IRCCS in Rome, will be included in the present study. Participants will be randomized into two groups: a Real group and a Sham group. Both groups will undergo a rehabilitation intervention using an immersive virtual reality system. The Real group will be exposed to scenarios containing specific stimuli for the visuo-vestibular system, while the Sham group will be exposed to the same scenarios but without specific stimuli. All participants in both groups will undergo 12 treatment sessions (three times a week), each lasting 20 minutes. All treatments will be conducted by physiotherapists specialized in neurological and vestibular rehabilitation. Patients will be assessed before the start of the treatment, at the end of the intervention, and one month after its completion, in order to evaluate the effects of the experimental training on balance and gait, and on the patient's perceived quality of life. Another aim will be to assess the user's satisfaction with the new proposed protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of hemorrhagic or ischemic stroke (more than 6 months from the acute event)
* Patients aged between 18 and 80 years
* Absence of cognitive deficits that may interfere with the patient's ability to understand the exercise instructions (MiniMentalState Evaluation > 24)
* Functional Ambulation Category ≥ 3
* Absence of associated orthopedic, visual, and/or neurological issues (clinically assessed) that may affect participation in the study

Exclusion Criteria:

* Patients with stroke (less than 6 months from the acute event);
* Patients aged under 18 and over 80;
* Presence of associated orthopedic, visual, and/or neurological issues (clinically assessed) that may affect participation in the study;
* Presence of cognitive deficits that may interfere with the patient's ability to understand the exercise instructions (MiniMentalState Evaluation ≤ 24);
* Epilepsy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Mini-BESTest | T0 (Baseline)
  The Mini-BESTest is a clinical scale used to assess balance and fall risk, consisting of 14 items covering anticipatory, reactive, dynamic balance, and transfers.
  Scoring: ranges from 0 (worst balance) to 28 (best balance); higher scores indicate better performance, while lower scores indicate greater fall risk or postural deficits.
Mini-BESTest | T1 (4 weeks from the baseline - end of treatment period)
  The Mini-BESTest is a clinical scale used to assess balance and fall risk, consisting of 14 items covering anticipatory, reactive, dynamic balance, and transfers.
  Scoring: ranges from 0 (worst balance) to 28 (best balance); higher scores indicate better performance, while lower scores indicate greater fall risk or postural deficits.
Mini-BESTest | T2 ( 4 weeks and 1 month from the baseline - 1 month follow up)
  The Mini-BESTest is a clinical scale used to assess balance and fall risk, consisting of 14 items covering anticipatory, reactive, dynamic balance, and transfers.
  Scoring: ranges from 0 (worst balance) to 28 (best balance); higher scores indicate better performance, while lower scores indicate greater fall risk or postural deficits.

SECONDARY OUTCOMES:
Berg Balance Scale | T0 (Baseline)
  The Berg Balance Scale (BBS) is a clinical tool used to assess static and dynamic balance through 14 functional tasks, such as standing, reaching, and turning.
  Scoring: ranges from 0 (poor balance) to 56 (excellent balance); higher scores indicate better balance, while lower scores suggest increased risk of falls.
Berg Balance Scale | T1 (4 weeks from the baseline - end of treatment period)
  The Berg Balance Scale (BBS) is a clinical tool used to assess static and dynamic balance through 14 functional tasks, such as standing, reaching, and turning.
  Scoring: ranges from 0 (poor balance) to 56 (excellent balance); higher scores indicate better balance, while lower scores suggest increased risk of falls.
Berg Balance Scale | T2 ( 4 weeks and 1 month from the baseline - 1 month follow up)
  The Berg Balance Scale (BBS) is a clinical tool used to assess static and dynamic balance through 14 functional tasks, such as standing, reaching, and turning.
  Scoring: ranges from 0 (poor balance) to 56 (excellent balance); higher scores indicate better balance, while lower scores suggest increased risk of falls.
Performance Oriented Mobility Assessment | T0 (Baseline)
  The Performance Oriented Mobility Assessment (POMA), also called the Tinetti Test, evaluates gait and balance to estimate fall risk in older adults. It includes two sections: balance (sitting, standing, turning) and gait (initiation, step length, symmetry).
  Scoring: total ranges from 0 (highest fall risk / worst performance) to 28 (lowest fall risk / best performance); higher scores indicate better mobility and lower fall risk.
Performance Oriented Mobility Assessment | T1 (4 weeks from the baseline - end of treatment period)
  The Performance Oriented Mobility Assessment (POMA), also called the Tinetti Test, evaluates gait and balance to estimate fall risk in older adults. It includes two sections: balance (sitting, standing, turning) and gait (initiation, step length, symmetry).
  Scoring: total ranges from 0 (highest fall risk / worst performance) to 28 (lowest fall risk / best performance); higher scores indicate better mobility and lower fall risk.
Performance Oriented Mobility Assessment | T2 ( 4 weeks and 1 month from the baseline - 1 month follow up)
  The Performance Oriented Mobility Assessment (POMA), also called the Tinetti Test, evaluates gait and balance to estimate fall risk in older adults. It includes two sections: balance (sitting, standing, turning) and gait (initiation, step length, symmetry).
  Scoring: total ranges from 0 (highest fall risk / worst performance) to 28 (lowest fall risk / best performance); higher scores indicate better mobility and lower fall risk.
Modified Barthel Index | T0 (Baseline)
  The Modified Barthel Index (MBI) is a scale that measures a person's independence in activities of daily living (ADLs), such as feeding, bathing, dressing, and mobility.
  Scoring: ranges from 0 (completely dependent) to 100 (completely independent); higher scores indicate greater independence, lower scores indicate more severe dependency.
Modified Barthel Index | T1 (4 weeks from the baseline - end of treatment period)
  The Modified Barthel Index (MBI) is a scale that measures a person's independence in activities of daily living (ADLs), such as feeding, bathing, dressing, and mobility.
  Scoring: ranges from 0 (completely dependent) to 100 (completely independent); higher scores indicate greater independence, lower scores indicate more severe dependency.
Modified Barthel Index | T2 ( 4 weeks and 1 month from the baseline - 1 month follow up)
  The Modified Barthel Index (MBI) is a scale that measures a person's independence in activities of daily living (ADLs), such as feeding, bathing, dressing, and mobility.
  Scoring: ranges from 0 (completely dependent) to 100 (completely independent); higher scores indicate greater independence, lower scores indicate more severe dependency.
Stroke Specific Quality of Life Scale | T0 (Baseline)
  The Stroke Specific Quality of Life Scale (SS-QOL) is a questionnaire designed to assess health-related quality of life in stroke survivors, covering physical, emotional, cognitive, and social domains.
  Scoring: total scores typically range from 49 (worst quality of life) to 245 (best quality of life), with higher scores reflecting better perceived well-being and function.
Stroke Specific Quality of Life Scale | T1 (4 weeks from the baseline - end of treatment period)
  The Stroke Specific Quality of Life Scale (SS-QOL) is a questionnaire designed to assess health-related quality of life in stroke survivors, covering physical, emotional, cognitive, and social domains.
  Scoring: total scores typically range from 49 (worst quality of life) to 245 (best quality of life), with higher scores reflecting better perceived well-being and function.
Stroke Specific Quality of Life Scale | T2 ( 4 weeks and 1 month from the baseline - 1 month follow up)
  The Stroke Specific Quality of Life Scale (SS-QOL) is a questionnaire designed to assess health-related quality of life in stroke survivors, covering physical, emotional, cognitive, and social domains.
  Scoring: total scores typically range from 49 (worst quality of life) to 245 (best quality of life), with higher scores reflecting better perceived well-being and function.
User Satisfaction Evaluation Questionnaire | T0 (Baseline)
  The User Satisfaction Evaluation Questionnaire (USEQ) is a tool used to measure users' satisfaction with a device, system, or service, focusing on usability, comfort, and overall experience.
  Scoring: typically ranges from 6 (lowest satisfaction) to 30 (highest satisfaction); higher scores indicate greater user satisfaction, while lower scores suggest issues or dissatisfaction.
User Satisfaction Evaluation Questionnaire | T1 (4 weeks from the baseline - end of treatment period)
  The User Satisfaction Evaluation Questionnaire (USEQ) is a tool used to measure users' satisfaction with a device, system, or service, focusing on usability, comfort, and overall experience.
  Scoring: typically ranges from 6 (lowest satisfaction) to 30 (highest satisfaction); higher scores indicate greater user satisfaction, while lower scores suggest issues or dissatisfaction.
User Satisfaction Evaluation Questionnaire | T2 ( 4 weeks and 1 month from the baseline - 1 month follow up)
  The User Satisfaction Evaluation Questionnaire (USEQ) is a tool used to measure users' satisfaction with a device, system, or service, focusing on usability, comfort, and overall experience.
  Scoring: typically ranges from 6 (lowest satisfaction) to 30 (highest satisfaction); higher scores indicate greater user satisfaction, while lower scores suggest issues or dissatisfaction.
Instrumental Gait Evaluation | T0 (Baseline)
  The instrumental motor assessment will be performed using seven wearable inertial sensors (128 Hz, Opal, APDM, Portland, Oregon, USA), which operate with an internal battery and are completely wireless. Each inertial sensor contains a triaxial accelerometer, capable of measuring accelerations along its three axes, which will align with the body axes (antero-posterior, lateral-lateral, cranio-caudal), and a triaxial gyroscope to measure angular velocities around these same axes. The seven wearable sensors will be placed using elastic supports at the level of the lambdoid suture of the skull, trunk, sacrum (L4-L5), tibias, and wrists. Accelerations and angular velocities of the body segments of interest will be measured, and from these, various parameters will be extrapolated both in the time and frequency domains. The motor assessment using inertial sensors will be conducted during the execution of four motor tasks: The 10 Meter Walk Test, The Fukuda Stepping Test, The Figure-of-8 Walk
Instrumental Gait Evaluation | T1 (4 weeks from the baseline - end of treatment period)
  The instrumental motor assessment will be performed using seven wearable inertial sensors (128 Hz, Opal, APDM, Portland, Oregon, USA), which operate with an internal battery and are completely wireless. Each inertial sensor contains a triaxial accelerometer, capable of measuring accelerations along its three axes, which will align with the body axes (antero-posterior, lateral-lateral, cranio-caudal), and a triaxial gyroscope to measure angular velocities around these same axes. The seven wearable sensors will be placed using elastic supports at the level of the lambdoid suture of the skull, trunk, sacrum (L4-L5), tibias, and wrists. Accelerations and angular velocities of the body segments of interest will be measured, and from these, various parameters will be extrapolated both in the time and frequency domains. The motor assessment using inertial sensors will be conducted during the execution of four motor tasks: The 10 Meter Walk Test, The Fukuda Stepping Test, The Figure-of-8 Walk
Instrumental Gait Evaluation | T2 ( 4 weeks and 1 month from the baseline - 1 month follow up)
  The instrumental motor assessment will be performed using seven wearable inertial sensors (128 Hz, Opal, APDM, Portland, Oregon, USA), which operate with an internal battery and are completely wireless. Each inertial sensor contains a triaxial accelerometer, capable of measuring accelerations along its three axes, which will align with the body axes (antero-posterior, lateral-lateral, cranio-caudal), and a triaxial gyroscope to measure angular velocities around these same axes. The seven wearable sensors will be placed using elastic supports at the level of the lambdoid suture of the skull, trunk, sacrum (L4-L5), tibias, and wrists. Accelerations and angular velocities of the body segments of interest will be measured, and from these, various parameters will be extrapolated both in the time and frequency domains. The motor assessment using inertial sensors will be conducted during the execution of four motor tasks: The 10 Meter Walk Test, The Fukuda Stepping Test, The Figure-of-8 Walk
Instrumental assessment of vestibular function | T0 (Baseline)
  The assessment of vestibular function will be performed using the Video Head Impulse Test, vHIT OtosuiteV®, GN Otometrics, Denmark. Data related to the gain of the vestibulo-ocular reflex (VOR) during the Head Impulse Paradigm (HIMP) and the Suppression Head Impulse Paradigm (SHIMP) will be considered.
Instrumental assessment of vestibular function | T1 (4 weeks from the baseline - end of treatment period)
  The assessment of vestibular function will be performed using the Video Head Impulse Test, vHIT OtosuiteV®, GN Otometrics, Denmark. Data related to the gain of the vestibulo-ocular reflex (VOR) during the Head Impulse Paradigm (HIMP) and the Suppression Head Impulse Paradigm (SHIMP) will be considered.
Instrumental assessment of vestibular function | T2 ( 4 weeks and 1 month from the baseline - 1 month follow up)
  The assessment of vestibular function will be performed using the Video Head Impulse Test, vHIT OtosuiteV®, GN Otometrics, Denmark. Data related to the gain of the vestibulo-ocular reflex (VOR) during the Head Impulse Paradigm (HIMP) and the Suppression Head Impulse Paradigm (SHIMP) will be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Jacopo Piermaria, Principal Investigator — Fondazione Santa Lucia IRCCS; Diego Piatti, PT, Study Chair — Fondazione Santa Lucia IRCCS; Sara De Angelis, MSc, Study Chair — Fondazione Santa Lucia IRCCS; Roberta Annicchiarico, MD, Study Chair — Fondazione Santa Lucia IRCCS; Matteo Marucci, PhD, Study Chair — Department of Psychology, Sapienza University of Rome, Rome, Italy; Laboratory of Neuroscience and Applied Technology, Santa Lucia Foundation IRCCS, Rome, Italy.; Viviana Betti, Prof., Study Chair — Department of Psychology, Sapienza University of Rome, Rome, Italy; Laboratory of Neuroscience and Applied Technology, Santa Lucia Foundation IRCCS, Rome, Italy.; Marco Tramontano, Prof, Study Director — Department of Biomedical and Neuromotor Sciences, University of Bologna, 40138 Bologna, Italy.; Unit of Occupational Medicine, IRCCS Azienda Ospedaliero-Universitaria di Bologna, 40138 Bologna, Italy
Locations (1):
- Fondazione Santa Lucia IRCCS, Roma, RM, Italy

REFERENCES:
- [Background] LeMarshall SJ, Stevens LM, Ragg NP, Barnes L, Foster J, Canetti EFD. Virtual reality-based interventions for the rehabilitation of vestibular and balance impairments post-concussion: a scoping review. J Neuroeng Rehabil. 2023 Mar 3;20(1):31. doi: 10.1186/s12984-023-01145-4. PMID 36869367
- [Background] Mao Y, Chen P, Li L, Huang D. Virtual reality training improves balance function. Neural Regen Res. 2014 Sep 1;9(17):1628-34. doi: 10.4103/1673-5374.141795. PMID 25368651
- [Background] Martino Cinnera A, Verna V, Marucci M, Tavernese A, Magnotti L, Matano A, D'Acunto C, Paolucci S, Morone G, Betti V, Tramontano M. Immersive Virtual Reality for Treatment of Unilateral Spatial Neglect via Eye-Tracking Biofeedback: RCT Protocol and Usability Testing. Brain Sci. 2024 Mar 15;14(3):283. doi: 10.3390/brainsci14030283. PMID 38539671
- [Background] Tramontano M, Russo V, Spitoni GF, Ciancarelli I, Paolucci S, Manzari L, Morone G. Efficacy of Vestibular Rehabilitation in Patients With Neurologic Disorders: A Systematic Review. Arch Phys Med Rehabil. 2021 Jul;102(7):1379-1389. doi: 10.1016/j.apmr.2020.11.017. Epub 2020 Dec 28. PMID 33383031